CLINICAL TRIAL: NCT05832437
Title: The Development and Pilot Testing of a Caregiver-Child Shared Decision-Making Intervention to Improve Asthma in Urban Youth
Brief Title: BREATHE-Peds Pilot- II III Trial and Post Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Maureen George, Professor of Nursing, Columbia University Irving Medical Center, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AAAT8015-Trial & Post-Trial; 1R21NR019668-01A1 (NIH)
Record Dates: First submitted 2023-04-10; First posted 2023-04-27 (Actual); Results first posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Asthma in Children
Keywords: Asthma; Adolescents; Dyads; Shared decision-making; Minority health
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient participants, data collectors, and the statistician will be blinded to assignment. Consent materials will inform patient participants that the focus of the trial is on the communication they have with their clinician about asthma management and control. Immediately after the intervention, patient participants will be asked to guess the condition to which their clinician had been randomized. At the end of participants' final data collection visit, data collectors will be asked to guess whether participants had received the active or control intervention at the visit. These data will provide some measurement of the success of masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BREATHE-Peds intervention (Experimental): The patient's primary care provider (PCP) will deliver a brief intervention using motivational interviewing and shared decision making, in a one time 9-minute intervention integrated into an office visit for asthma. PCPs will follow a 4-step script tailored to erroneous asthma and inhaled corticosteroid (ICS) beliefs, as well as ACQ score, measured just prior to the office visit.
  Interventions: Behavioral: BREATHE-Peds Intervention
- Control Intervention (Active Comparator): The patient's primary care provider (PCP) will deliver a 9-minute scripted intervention on credible nutrition and lifestyle information. The control intervention is designed to not be specific enough to change strategies related to asthma control.
  Interventions: Behavioral: Control Intervention

INTERVENTIONS:
Behavioral: BREATHE-Peds Intervention — BREATHE-Peds utilizes Primary Care Providers (PCPs) to deliver a 4-step script that was created by and tailored to Black adults' asthma and inhaled corticosteroid beliefs, as well as their Asthma Control Questionnaire (ACQ) score, measured just prior to the medical visit. Step 1: Raise the subject (1½ minute). Step 2: Provide feedback (1½ minutes). Step 3: Enhance engagement (3 minutes). Step 4: Shared decision-making (3 minutes).
  Arms: BREATHE-Peds intervention
Behavioral: Control Intervention — The control intervention will be a 9-minute scripted discussion tailored to living a health lifestyle. Step 1: Review of BMI, current diet and exercise (3 minutes). Step 2: Diet/exercise counseling (3 minutes). Step 3: Plan for goal attainment (3 minutes).
  Arms: Control Intervention

SUMMARY:
The overall aims of this study are to develop and pilot test BRief intervention to Evaluate Asthma THErapy (BREATHE)-Peds, a dyadic shared decision-making intervention, to improve asthma by supporting self-management among racial and ethnic minority early adolescents receiving care for uncontrolled asthma in federally-qualified health centers (FQHCs) in urban communities. Aim 1 (Phase I) involves developing the intervention through focus groups with early adolescents and caregivers. Aims 2 and 3 (Phase II) involve preliminary testing of the intervention through a pilot randomized controlled trial. This record is for Phase II and III only

DETAILED DESCRIPTION:
Despite high asthma prevalence and morbidity among adolescents (highest among Black and Hispanic youth and early adolescents aged 10-14), there is a lack of developmentally appropriate interventions for this at-risk group. Racial and ethnic minority early adolescents have sub-optimal asthma self-management. Critical health behaviors that emerge during early adolescence affect lifelong patterns; therefore, early adolescence offers a unique opportunity to intervene. Additionally, successful self-management requires the right division of responsibility between adolescents and their caregivers. Thus, intervening simultaneously with early adolescents and their caregivers who can help support the adolescent's growing autonomy to self-manage their condition has the potential for a synergistic effect.

Prior studies have demonstrated the effects of improved asthma control of BREATHE, a brief one-time shared decision-making intervention for Black adults with uncontrolled asthma that utilizes motivational interviewing delivered by primary care providers. This study (i.e., Phase II and Phase III) ) a pilot validation phase will conduct a group-randomized trial in two FQHCs with 85 dyads treated by 8 PCPs (10 dyads/PCP) randomized to 1 of 2 study arms: (a) BREATHE-PEDS-Peds (n=42 dyads), or (b) dose-matched attention control (n=43 dyads). Post-trial interviews with PCPs, caregivers, and their children to evaluate satisfaction with the intervention will be conducted; caregiver-child dyads will be followed for 3 months post-intervention to assess the impact of BREATHE-PEDS-Peds on asthma outcomes.

ELIGIBILITY:
Inclusion Criteria (Dyad participants):

Dyad (caregiver/child) participants will

1. Early adolescents (10-14 years of age) or the caregiver of early adolescents (10-14 years of age)
2. Have or the caregiver of a child that has clinician-diagnosed persistent asthma (defined as being prescribed inhaled corticosteroids in the last 12 months)
3. Receive asthma care at a partner FQHC and
4. Child screens positive for uncontrolled asthma as measured by the Asthma Control Questionnaire- 6 items (ACQ-6) and child or caregiver has erroneous beliefs as measured by the Conventional and Alternative Management for Asthma (CAM-A) survey.

Inclusion Criterion (clinicians):

1. Those who manage a panel of pediatric asthma patients at partner FQHC.

Exclusion Criteria (Dyad participants):

1. Non-English speaking
2. Serious mental health conditions that preclude completion of study procedures or confound analyses or participation in a listening session

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen George, PhD, Principal Investigator — Columbia University; Jean-Marie Bruzzese, PhD, Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - Urban Health Plan: Adolescent Health and Wellness, The Bronx, New York
  - Urban Health Plan: El Nuevo San Juan, The Bronx, New York
  - Urban Health Plan: Bella Vista, The Bronx, New York

REFERENCES:
- [Background] Centers for Disease Control. Asthma Surveillance Data. Retrieved from https://www.cdc.gov/asthma/asthmadata.htm October 20, 2020.
- [Background] Zahran HS, Bailey CM, Damon SA, Garbe PL, Breysse PN. Vital Signs: Asthma in Children - United States, 2001-2016. MMWR Morb Mortal Wkly Rep. 2018 Feb 9;67(5):149-155. doi: 10.15585/mmwr.mm6705e1. PMID 29420459
- [Background] Akinbami LJ, Moorman JE, Garbe PL, Sondik EJ. Status of childhood asthma in the United States, 1980-2007. Pediatrics. 2009 Mar;123 Suppl 3:S131-45. doi: 10.1542/peds.2008-2233C. PMID 19221156
- [Background] Claudio L, Stingone JA, Godbold J. Prevalence of childhood asthma in urban communities: the impact of ethnicity and income. Ann Epidemiol. 2006 May;16(5):332-40. doi: 10.1016/j.annepidem.2005.06.046. Epub 2005 Oct 20. PMID 16242960
- [Background] Lara M, Akinbami L, Flores G, Morgenstern H. Heterogeneity of childhood asthma among Hispanic children: Puerto Rican children bear a disproportionate burden. Pediatrics. 2006 Jan;117(1):43-53. doi: 10.1542/peds.2004-1714. PMID 16396859
- [Background] Bruzzese JM, Bonner S, Vincent EJ, Sheares BJ, Mellins RB, Levison MJ, Wiesemann S, Du Y, Zimmerman BJ, Evans D. Asthma education: the adolescent experience. Patient Educ Couns. 2004 Dec;55(3):396-406. doi: 10.1016/j.pec.2003.04.009. PMID 15582346
- [Background] Dahl RE, Allen NB, Wilbrecht L, Suleiman AB. Importance of investing in adolescence from a developmental science perspective. Nature. 2018 Feb 21;554(7693):441-450. doi: 10.1038/nature25770. PMID 29469094
- [Background] Williams PG, Holmbeck GN, Greenley RN. Adolescent health psychology. J Consult Clin Psychol. 2002 Jun;70(3):828-42. PMID 12090386
- [Background] Maggs JL, Schulenberg J, Hurrelmann K. Developmental transitions during adolescence: health promotion implications. In: Schulenberg J, Maggs JL, Hurrelman K, eds. Health Risks and Developmental Transitions During Adolescence. New York: Cambridge University Press. 1997;522-546.
- [Background] Klok T, Kaptein AA, Brand PLP. Non-adherence in children with asthma reviewed: The need for improvement of asthma care and medical education. Pediatr Allergy Immunol. 2015 May;26(3):197-205. doi: 10.1111/pai.12362. PMID 25704083
- [Background] Rhee H, Belyea MJ, Brasch J. Family support and asthma outcomes in adolescents: barriers to adherence as a mediator. J Adolesc Health. 2010 Nov;47(5):472-8. doi: 10.1016/j.jadohealth.2010.03.009. Epub 2010 May 14. PMID 20970082
- [Background] Yang TO, Sylva K, Lunt I. Parent support, peer support, and peer acceptance in healthy lifestyle for asthma management among early adolescents. J Spec Pediatr Nurs. 2010 Oct;15(4):272-81. doi: 10.1111/j.1744-6155.2010.00247.x. PMID 20880275
- [Background] Bruzzese JM, Stepney C, Fiorino EK, Bornstein L, Wang J, Petkova E, Evans D. Asthma self-management is sub-optimal in urban Hispanic and African American/black early adolescents with uncontrolled persistent asthma. J Asthma. 2012 Feb;49(1):90-7. doi: 10.3109/02770903.2011.637595. Epub 2011 Dec 7. PMID 22149141
- [Background] Holley S, Morris R, Knibb R, Latter S, Liossi C, Mitchell F, Roberts G. Barriers and facilitators to asthma self-management in adolescents: A systematic review of qualitative and quantitative studies. Pediatr Pulmonol. 2017 Apr;52(4):430-442. doi: 10.1002/ppul.23556. Epub 2016 Oct 7. PMID 27717193
- [Background] Bruzzese JM, Unikel L, Gallagher R, Evans D, Colland V. Feasibility and impact of a school-based intervention for families of urban adolescents with asthma: results from a randomized pilot trial. Fam Process. 2008 Mar;47(1):95-113. doi: 10.1111/j.1545-5300.2008.00241.x. PMID 18411832
- [Background] George M, Bruzzese JM, Lynn S Sommers M, Pantalon MV, Jia H, Rhodes J, Norful AA, Chung A, Chittams J, Coleman D, Glanz K. Group-randomized trial of tailored brief shared decision-making to improve asthma control in urban black adults. J Adv Nurs. 2021 Mar;77(3):1501-1517. doi: 10.1111/jan.14646. Epub 2020 Nov 29. PMID 33249632

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 30 dyads (30 pediatric patients + 30 caregivers) were randomized to the intervention and 30 dyads (30 pediatric patients + 30 caregivers) were randomized to the control group.
Groups:
- BREATHE-Peds Intervention (PCPs): Providers which delivered the intervention were considered participants.
- BREATHE-Peds Intervention (Dyads): The patient's primary care provider (PCP) will deliver a brief intervention using motivational interviewing and shared decision making, in a one time 9-minute intervention integrated into an office visit for asthma. PCPs will follow a 4-step script tailored to erroneous asthma and inhaled corticosteroid (ICS) beliefs, as well as ACQ score, measured just prior to the office visit. PCPs will follow a 4-step script tailored to erroneous asthma and inhaled corticosteroid (ICS) beliefs, as well as ACQ score, measured just prior to the office visit.
  BREATHE-Peds Intervention: BREATHE-Peds utilizes Primary Care Providers (PCPs) to deliver a 4-step script that was created by and tailored to Black adults' asthma and inhaled corticosteroid beliefs, as well as their Asthma Control Questionnaire (ACQ) score, measured just prior to the medical visit. Step 1: Raise the subject (1½ minute). Step 2: Provide feedback (1½ minutes). Step 3: Enhance engagement (3 minutes). Step 4: Shared decision-making (3 minutes).
- Control Intervention (PCPs): Providers which delivered the control intervention were considered participants.
- Control Intervention (Dyads): The patient's primary care provider (PCP) will deliver a 9-minute scripted intervention on credible nutrition and lifestyle information. The control intervention is designed to not be specific enough to change strategies related to asthma control.
  Control Intervention: The control intervention will be a 9-minute scripted discussion tailored to living a health lifestyle. Step 1: Review of BMI, current diet and exercise (3 minutes). Step 2: Diet/exercise counseling (3 minutes). Step 3: Plan for goal attainment (3 minutes).
Period: Overall Study
Arm/Group | BREATHE-Peds Intervention (PCPs) | BREATHE-Peds Intervention (Dyads) | Control Intervention (PCPs) | Control Intervention (Dyads)
Started | 3 | 30 (30 Dyads (60 Unique individuals: 30 caregivers + 30 pediatric patients)) | 4 | 30 (30 Dyads (60 Unique individuals: 30 caregivers + 30 pediatric patients))
Completed | 2 | 30 (30 Dyads (60 Unique individuals: 30 caregivers + 30 pediatric patients)) | 4 | 30 (30 Dyads (60 Unique individuals: 30 caregivers + 30 pediatric patients))
Not Completed | 1 | 0 | 0 | 0
Not completed — time off work | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data was collected for the PCPs, and pediatric patients and their caregivers.
Groups:
- BREATHE-Peds Intervention (Child in Dyads); BREATHE-Peds Intervention (Caregiver in Dyads): The patient's primary care provider (PCP) will deliver a brief intervention using motivational interviewing and shared decision making, in a one time 9-minute intervention integrated into an office visit for asthma. PCPs will follow a 4-step script tailored to erroneous asthma and inhaled corticosteroid (ICS) beliefs, as well as ACQ score, measured just prior to the office visit. PCPs will follow a 4-step script tailored to erroneous asthma and inhaled corticosteroid (ICS) beliefs, as well as ACQ score, measured just prior to the office visit.
  BREATHE-Peds Intervention: BREATHE-Peds utilizes Primary Care Providers (PCPs) to deliver a 4-step script that was created by and tailored to Black adults' asthma and inhaled corticosteroid beliefs, as well as their Asthma Control Questionnaire (ACQ) score, measured just prior to the medical visit. Step 1: Raise the subject (1½ minute). Step 2: Provide feedback (1½ minutes). Step 3: Enhance engagement (3 minutes). Step 4: Shared decision-making (3 minutes).
- Control Intervention (Child in Dyads); Control Intervention (Caregivers in Dyad): The patient's primary care provider (PCP) will deliver a 9-minute scripted intervention on credible nutrition and lifestyle information. The control intervention is designed to not be specific enough to change strategies related to asthma control.
  Control Intervention: The control intervention will be a 9-minute scripted discussion tailored to living a health lifestyle. Step 1: Review of BMI, current diet and exercise (3 minutes). Step 2: Diet/exercise counseling (3 minutes). Step 3: Plan for goal attainment (3 minutes).
- Total: Total of all reporting groups
Arm/Group | BREATHE-Peds Intervention (PCPs) | BREATHE-Peds Intervention (Child in Dyads) | BREATHE-Peds Intervention (Caregiver in Dyads) | Control Intervention (PCPs) | Control Intervention (Child in Dyads) | Control Intervention (Caregivers in Dyad) | Total
Number analyzed (Participants) | 3 | 30 | 30 | 4 | 30 | 30 | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 30 | 0 | 0 | 30 | 0 | 60
  Between 18 and 65 years | 2 | 0 | 29 | 4 | 0 | 30 | 65
  >=65 years | 1 | 0 | 1 | 0 | 0 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.33 (13.50) | 11.3 (0.99) | 39.43 (8.92) | 43.75 (13.64) | 11.1 (0.92) | 36.86 (6.45) | 15.03 (12.03)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant in control group did not report sex.
  Participants
    number analyzed (Participants) | 3 | 30 | 30 | 4 | 29 | 30 | 126
    Female | 2 | 16 | 27 | 4 | 13 | 29 | 91
    Male | 1 | 14 | 3 | 0 | 16 | 1 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 23 | 23 | 1 | 27 | 27 | 102
  Not Hispanic or Latino | 2 | 6 | 6 | 3 | 3 | 3 | 23
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 8 | 7 | 3 | 4 | 6 | 28
  White | 1 | 1 | 1 | 0 | 0 | 0 | 3
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 21 | 22 | 0 | 26 | 24 | 93

OUTCOME MEASURES:

1. Primary Outcome: Mean Asthma Control Questionnaire Score
Description: Asthma control as measured by improvements in Asthma Control Questionnaire (ACQ) score, a 6-item validated and widely used measure of asthma control. Each question is rated from 0 to 6. A score of 0 indicates well controlled asthma and a score of 6 indicates extremely poorly controlled asthma. The overall ACQ score is the mean score of all 6 items with scores ranging from 0 to 6. Lower mean scores indicate greater asthma control (better outcome), higher mean scores indicate lesser asthma control.
Time Frame: Up to 3 months post intervention
Population: Pediatric patient participants only
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- BREATHE-Peds Intervention: The patient's primary care provider (PCP) will deliver a brief intervention using motivational interviewing and shared decision making, in a one time 9-minute intervention integrated into an office visit for asthma. PCPs will follow a 4-step script tailored to erroneous asthma and inhaled corticosteroid (ICS) beliefs, as well as ACQ score, measured just prior to the office visit. PCPs will follow a 4-step script tailored to erroneous asthma and inhaled corticosteroid (ICS) beliefs, as well as ACQ score, measured just prior to the office visit.
  BREATHE-Peds Intervention: BREATHE-Peds utilizes Primary Care Providers (PCPs) to deliver a 4-step script that was created by and tailored to Black adults' asthma and inhaled corticosteroid beliefs, as well as their Asthma Control Questionnaire (ACQ) score, measured just prior to the medical visit. Step 1: Raise the subject (1½ minute). Step 2: Provide feedback (1½ minutes). Step 3: Enhance engagement (3 minutes). Step 4: Shared decision-making (3 minutes).
Arm/Group | BREATHE-Peds Intervention | Control Intervention
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline | 2.7 (0.57) | 2.63 (0.62)
  Month 1 | 0.98 (0.98) | 0.82 (0.79)
  Month 2 | 0.80 (0.85) | 0.58 (0.64)
  Month 3 | 0.95 (1.05) | 0.68 (0.76)

2. Secondary Outcome: Mean Shared Decision Making-Questionnaire-9 Score
Description: The Shared Decision Making (SDM) Questionnaire-9, is a patient reported, 9-item validated instrument that consists of nine statements that measure the decisional process in medical visits from both patients' and physicians' perspectives. Each statement is rated on a six-point scale from "completely disagree" (0) to "completely agree" (5). The raw total score of all items range from 0-45. Lower scores indicate lower levels of shared decision making between provider and patient (in this study as it pertains to asthma treatment) and higher scores indicate higher levels of shared decision making (better outcome).
Time Frame: Baseline (immediately post-intervention)
Population: Pediatric patient participants only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BREATHE-Peds Intervention | Control Intervention
Number analyzed (Participants) | 30 | 29
score on a scale | 42.9 (8.10) | 39.55 (8.89)

3. Secondary Outcome: Mean Medication Adherence Report Scale - Asthma Score
Description: Inhaled corticosteroid adherence as measured by the Medication Adherence Report Scale - Asthma (MARS-A). Participants are asked to rate the frequency with which they engage in each of the adherence-related behaviors on a five-point scale, where 5 = never, 4 = rarely, 3 = sometimes, 2 = often and 1 = always. Scores for each item are summed to give a total score ranging from 1 to 5, with higher scores indicating higher levels of reported adherence.
Time Frame: Up to 3 months post intervention
Population: Pediatric patient participants who were prescribed ICS at baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BREATHE-Peds Intervention | Control Intervention
Number analyzed (Participants) | 23 | 20
score on a scale
  Baseline | 4.13 (0.81) | 3.87 (0.80)
  Month 1 | 4.13 (0.88) | 4.05 (0.77)
  Month 2 | 4.34 (0.68) | 4.26 (0.87)
  Month 3 | 4.45 (0.683) | 4.48 (0.73)

4. Secondary Outcome: Mean Asthma Quality of Life Questionnaire Score
Description: Asthma quality of life improvements as measured by the Asthma Quality of Life Questionnaire (AQLQ), a 32-item validated and widely-used measure consisting of 4 domains: symptoms (11 items), emotions (5 items), environment (4 items), and activities (12 items). Each item is measured on a 7-point Likert scale (7 = not impaired at all, 1 = severely impaired). The overall AQLQ score is the mean of all 32 responses and the individual domain scores are the means of the items in those domains. The overall score ranges from 1 to 7, where lower mean scores indicate lower quality of life due to asthma (worse outcome).
Time Frame: Up to 3 months post intervention
Population: Pediatric patient participants only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BREATHE-Peds Intervention | Control Intervention
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline | 5.37 (1.32) | 5.72 (1.05)
  Month 1 | 5.78 (1.24) | 6.44 (0.80)
  Month 3 | 5.89 (1.19) | 6.17 (1.21)

5. Secondary Outcome: Mean Asthma Impairment and Risk Questionnaire Score
Description: Asthma Impairment and Risk Questionnaire (AIRQ) is a 10-item valid and reliable survey that measures bot domains of control: symptom impairments and risk for uncontrolled asthma. AIRQ™ score ranges from 0-10, measured by total number of YES answers. Score tally of 0-1 indicates well controlled asthma, scores 2-4 indicate not well controlled asthma, and scores 5-10 indicate very poorly controlled asthma.
Time Frame: Up to 3 months post intervention
Population: Pediatric patient participants 12 years of age and older
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BREATHE-Peds Intervention | Control Intervention
Number analyzed (Participants) | 14 | 11
score on a scale
  Baseline | 2.79 (2.55) | 3.00 (2.10)
  Month 1 | 1.46 (1.98) | 1.64 (2.46)
  Month 2 | 1.08 (1.31) | 1.45 (2.21)
  Month 3 | 1.75 (1.71) | 1.82 (1.94)

ADVERSE EVENTS:
Time Frame: 3 months
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed for the Clinicians or Caregiver participants.
Arm/Group | BREATHE-Peds Intervention (PCPs) | BREATHE-Peds Intervention (Dyads) | Control Intervention (Dyads) | Control Intervention (PCPs)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/30 | 0/30 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/30 | 0/30 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/30 | 0/30 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT05832437/Prot_SAP_000.pdf